CLINICAL TRIAL: NCT02860104
Title: Ultrasound Guided Percutaneous Microwave Ablation for Breast Lesions: A Prospective Multicenter Study
Brief Title: Ultrasound Guided Percutaneous Microwave Ablation for Breast Lesions
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chair, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 939530lp
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasm of Breast
Keywords: microwave ablation; breast; multicenter
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- microwave ablation (Other): microwave ablation
  Interventions: Device: microwave ablation

INTERVENTIONS:
Device: microwave ablation — ultrasound guided percutaneous microwave ablation for breast lesions

SUMMARY:
The investigators will perform this study to prospectively analyse the clinical outcome after percutaneous microwave ablation(MWA) of benign and malignant breast lesion under ultrasound (US) guidance.

DETAILED DESCRIPTION:
A total of more than 500 patients diagnosed with benign breast lesions and 50 patients with malignant breast lesions in seven centers of China will be recruited in this study and underwent US-guided percutaneous MWA treatment. Information for each patient includes demographics; longest diameters of tumors; tumor numbers; tumor pathological type; location of tumor according to whether adjacent to skin, pectoralis, areola and papilla. Ablation variables including session, puncture, time, and power; complete ablation, complications; reduction in volume, palpability, pain and cosmetic satisfying outcomes,recurrence,survival will be measured and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* breast lesion proved by using core-needle biopsy;
* for benign lesions,lesion 1.0 cm or larger in greatest diameter and continually increasing during a half year follow-up; for malignant ones, lesion size 2cm or smaller;
* distance of at least 1.0cm to papilla with the patients supine;
* the symptoms of local pain, discomfortable or compression considered probably relating to the lesion of breast;
* the patient with evidently psychological pressure due to the occurrence of the lesion;
* patients unwilling or refused to receive other treatment and presence of an appropriate route for percutaneous puncture under US guidance.

Exclusion Criteria:

* patients who were pregnant or breast-feeding;
* patients with evidence of coagulopathy or acute or severe pulmonary insufficiency or heart dysfunction;
* patients during menstrual period;
* patients who wanted to undergo other therapies including surgical excision and vacuum-assisted biopsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
reduction in volume | 5 year
  the volume reduction ratio (VRR) which was calculated by the following equation: VRR (%) = [(initial volume - final volume) × 100]/initial volume.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
cosmetics effect, volume reduction rate,complications

REFERENCES:
- [Derived] Yang Q, Li H, Chen BH, He GZ, Wu XP, Wang LX, Wu H, Dou JP, Han ZY, Zhang J, Yu XL, Yu J, Liang P. Ultrasound-guided percutaneous microwave ablation for 755 benign breast lesions: a prospective multicenter study. Eur Radiol. 2020 Sep;30(9):5029-5038. doi: 10.1007/s00330-020-06868-9. Epub 2020 Apr 30. PMID 32356159
- [Derived] Yu J, Wu H, Meng XW, Mu MJ, Dou JP, Ahmed M, Liang P. Ultrasound-guided percutaneous microwave ablation of central intraductal papilloma: a prospective pilot study. Int J Hyperthermia. 2019;36(1):606-612. doi: 10.1080/02656736.2019.1619849. PMID 31179781